CLINICAL TRIAL: NCT02437721
Title: Suitability of an Infant Formula With L-5-Methyltetrahydrofolate for the Particular Nutritional Use in Infants
Acronym: MEFOLIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: University Clinic Dr Dragisa Misovic-Dedinje (Other); HiPP GmbH & Co. Vertrieb KG (Industry); Institute for Laboratory Diagnostics Konzilijum (Unknown); Bevital AS (Unknown); Charite University, Berlin, Germany (Other); Sermon CRO (Industry); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2014-05-06-MTHF
Record Dates: First submitted 2015-03-30; First posted 2015-05-08 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-01

CONDITIONS: Growth and Development
MeSH Terms: interventions — Folic Acid; 5-methyltetrahydrofolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- infant formula containing folic acid (Active Comparator): Infant formula including folic acid within the range stipulated by European legislation on infant formula
  Interventions: Other: infant formula containing folic acid
- infant formula containing MTHF (Experimental): Infant formula including MTHF instead of folic acid
  Interventions: Other: infant formula containing MTHF
- Breast milk (No Intervention): non randomized reference group

INTERVENTIONS:
Other: infant formula containing folic acid
  Other Names: folic acid
  Arms: infant formula containing folic acid
Other: infant formula containing MTHF
  Other Names: L-5-Methyltetrahydrofolate
  Arms: infant formula containing MTHF

SUMMARY:
The study is designed to show equivalence of an infant formula containing L-5- Methyltetrahydrofolate (MTHF) compared to a standard infant formula containing folic acid in respect to weight gain of healthy term infants receiving these infant formulae exclusively during the first 4 months of life. Healthy non breast fed infants will be randomized to receive either a standard infant formula with folic acid or a corresponding formula with MTHF instead of folic acid. Besides weight and length further anthropometric measures will be taken monthly from the age of 4 weeks to the age of 16 weeks and at the age 4 and 16 weeks blood samples will be taken for the determination of folate status and genotyping. As a reference the same measures will be taken in a group of breast fed infants, whose mothers' folate status will be determined as well.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (by parents, caregiver)
* Healthy male or female infants <28 days of life
* Gestational age at delivery ≥37 and ≤42 weeks
* Birth weight between 2500 - 4500g
* Parents / Caregivers are able to speak Serbian language

Exclusion Criteria:

* Serious acquired or congenital diseases that is expected to interfere with normal feeding or growth
* Feeding of more than 10% of energy (1 bottle/day) from sources other than the formula (or breast milk in the reference group) at inclusion
* Participation in another clinical study
* Mothers with diabetes mellitus (including gestational diabetes)
* Reason to presume that the parents are unable to meet the study plan requirements
* Diseases of the mother which have an effect on the child's gastro-intestinal tract/ability to be fed
* Major abnormalities in hematological parameters
* Major abnormalities in hepatic, renal or metabolic functions
* Use of medication and vitamin supplements except vitamin K or D supplementation or vaccination
* Mother follows a vegan diet

Ages: 1 Day to 27 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2015-05; Primary Completion 2017-08 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
weight gain (gram/day) | age of 4 weeks until age of 16 weeks

SECONDARY OUTCOMES:
body length gain (cm/day) | age of 4 weeks until age of 16 weeks
fronto-occipital head circumference gain (in cm/day) | at age of 4 weeks and at the age of 16 weeks
dietary intake of study formula, non-study formula, additional liquids and solids | during the period age 4 weeks to age 16 weeks
  dietary intake will be determined as kcal per day and as kcal per kg body weight per day
feeding related behavior questionnaire | during the period age 4 weeks to age 16 weeks
stool characteristics (color and consistency) | during the period age 4 weeks to age 16 weeks
  stool characteristics are assessed by the Bristol scale criteria

OTHER OUTCOMES:
plasma levels of 5-MTHF in infants | at age of 4 weeks and at the age of 16 weeks
plasma levels of folic acid in infants | at age of 4 weeks and at the age of 16 weeks
plasma levels of 5-Formyl-tetrahydrofolate (fTHF) in infants | at age of 4 weeks and at the age of 16 weeks
plasma levels of 4-Alfa-hydroxy-5-methyl-THF (hmTHF) in infants | at age of 4 weeks and at the age of 16 weeks
plasma levels of Para-aminobenzoylglutamate (pABG) in infants | at age of 4 weeks and at the age of 16 weeks
plasma levels of Acetamidobenzoylglutamate (apABG) in infants | at age of 4 weeks and at the age of 16 weeks
red cell total folate in infants | at age of 4 weeks and at the age of 16 weeks
plasma levels of 5-MTHF in breast feeding mothers | at the infantile age of 8 weeks
breast milk levels of 5-MTHF in breast feeding mothers | at the infantile age of 8 weeks
plasma levels of folic acid in breast feeding mothers | at the infantile age of 8 weeks
breast milk levels of folic acid in breast feeding mothers | at the infantile age of 8 weeks
plasma levels of fTHF in breast feeding mothers | at the infantile age of 8 weeks
breast milk levels of fTHF in breast feeding mothers | at the infantile age of 8 weeks
plasma levels of hmTHF in breast feeding mothers | at the infantile age of 8 weeks
breast milk levels of hmTHF in breast feeding mothers | at the infantile age of 8 weeks
plasma levels of pABG in breast feeding mothers | at the infantile age of 8 weeks
breast milk levels of pABG in breast feeding mothers | at the infantile age of 8 weeks
plasma levels of apABG in breast feeding mothers | at the infantile age of 8 weeks
breast milk levels of apABG in breast feeding mothers | at the infantile age of 8 weeks
hemoglobin value of the breast feeding mothers | at the infantile age of 8 weeks
hematocrit value of the breast feeding mothers | at the infantile age of 8 weeks
mean corpuscular volume (MCV) of the breast feeding mothers | at the infantile age of 8 weeks
weight of infants | at infantile age 1 year
length of infants | at infantile age 1 year
head circumference of infants | at infantile age 1 year
hemoglobin value of infants | between Day 1 and Day 27 of life, at infantile age of 16 weeks and of 12 months
hematocrit value of infants | between Day 1 and Day 27 of life, at infantile age of 16 weeks and of 12 months
mean corpuscular volume (MCV) of infants | between Day 1 and Day 27 of life, at infantile age of 16 weeks and of 12 months
infantile genotype of methylenetetrahydrofolate-reductase | at infantile age 4 weeks
intake of folic acid in breast feeding mothers | at the infantile age of 8 weeks
intake of MTHF in breast feeding mothers | at the infantile age of 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, Prof., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (2):
- Serbia (2):
  - KBC Dr Dragiša Mišović-Dedinje, Belgrade
  - HiPP Clinical Study Center, Belgrade

REFERENCES:
- [Derived] Obeid R, Warnke I, Wittke A, Bendik I, Troesch B, Schoop R, Hecht C, Demmelmair J, Koletzko B; MEFOLIN Study Group. Infant blood concentrations of folate markers and catabolites are modified by 5,10-methylenetetrahydrofolate reductase C677T genotype and dietary folate source. Am J Clin Nutr. 2023 Mar;117(3):509-517. doi: 10.1016/j.ajcnut.2022.09.002. PMID 36872017
- [Derived] Troesch B, Demmelmair J, Gimpfl M, Hecht C, Lakovic G, Roehle R, Sipka L, Trisic B, Vusurovic M, Schoop R, Zdjelar S, Koletzko B; MEFOLIN Study Group. Suitability and safety of L-5-methyltetrahydrofolate as a folate source in infant formula: A randomized-controlled trial. PLoS One. 2019 Aug 19;14(8):e0216790. doi: 10.1371/journal.pone.0216790. eCollection 2019. PMID 31425504